CLINICAL TRIAL: NCT05542823
Title: Effect of Cuff Pressure of Endotracheal Tube on Postoperative Sore Throat: a Prospective Observational Study
Brief Title: Effect of Cuff Pressure of Endotracheal Tube on POST
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyun-Kyu Yoon, Clinical assistant professor, Seoul National University Hospital
Other Study IDs: POST_cuff_pressure
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Laparoscopic Surgery; Tracheal Intubation Morbidity; Sore-throat
Keywords: Laparoscopic surgery; Endotracheal intubation; Cuff pressure; Sore throat; Hoarseness
MeSH Terms: conditions — Pharyngitis; Hoarseness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this study is to evaluate the association between the duration of intraoperative cuff overpressure and the development of postoperative sore throat.

DETAILED DESCRIPTION:
For patients undergoing laparoscopic surgery after tracheal intubation, continuous cuff pressure monitoring is performed by connecting a pressure monitor to the cuff of the endotracheal tube. The incidence of postoperative sore throat was evaluated via direct questioning in all patients. This study aimed to investigate the association between the development of postoperative sore throat and the duration of overpressure in the cuff of the endotracheal tube.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing laparoscopic surgery and endotracheal intubation under general anesthesia

Exclusion Criteria:

* Patients who already had sore throat and hoarseness before surgery
* Patients who were expected to have anticipated difficult airway
* Surgery duration < 1 hour

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing laparoscopic surgery and endotracheal intubation under general anesthesia
Sampling Method: Probability Sample
Enrollment: 337 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2025-08-07 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative sore throat at 24h postoperatively. | at 24h postoperatively.
  Incidence of postoperative sore throat (score 1 or more) 0 = no sore throat
  1. = mild sore throat (less severe 1 = mild sore throat (less severe than with a cold)
  2. = moderate sore throat (as with a cold)2 = moderate sore throat (as with a cold)
  3. = severe (more severe than with a cold)3 = severe (more severe than with a cold)

SECONDARY OUTCOMES:
Incidence of postoperative sore throat at 1h postoperatively. | at 1h postoperatively
  Incidence of postoperative sore throat (score 1 or more) 0 = no sore throat
  1. = mild sore throat (less severe 1 = mild sore throat (less severe than with a cold)
  2. = moderate sore throat (as with a cold)2 = moderate sore throat (as with a cold)
  3. = severe (more severe than with a cold)3 = severe (more severe than with a cold)
Incidence of postoperative sore throat at 48h postoperatively. | at 48h postoperatively
  Incidence of postoperative sore throat (score 1 or more) 0 = no sore throat
  1. = mild sore throat (less severe 1 = mild sore throat (less severe than with a cold)
  2. = moderate sore throat (as with a cold)2 = moderate sore throat (as with a cold)
  3. = severe (more severe than with a cold)3 = severe (more severe than with a cold)
Incidence of postoperative hoarseness at 1h postoperatively. | at 1h postoperatively
  Incidence of postoperative hoarseness (score 1 or more) 0 = no hoarseness
  1. = mild hoarseness (noticed by the patient only)
  2. = severe hoarseness (noticed by the time of the interview by the personnel)
  3. = aphonia (inability to speak)
Incidence of postoperative hoarseness at 24h postoperatively. | at 24h postoperatively.
  Incidence of postoperative hoarseness (score 1 or more) 0 = no hoarseness
  1. = mild hoarseness (noticed by the patient only)
  2. = severe hoarseness (noticed by the time of the interview by the personnel)
  3. = aphonia (inability to speak)
Incidence of postoperative hoarseness at 48h postoperatively. | at 48h postoperatively
  Incidence of postoperative hoarseness (score 1 or more) 0 = no hoarseness
  1. = mild hoarseness (noticed by the patient only)
  2. = severe hoarseness (noticed by the time of the interview by the personnel)
  3. = aphonia (inability to speak)

CONTACTS AND LOCATIONS:
Overall Officials: Hyun-Kyu Yoon, Principal Investigator — Seoul National University
Locations (2):
- South Korea (2):
  - Seoul national university hospital, Seoul, Please Select An Option
  - Hyun-Kyu Yoon, Seoul